CLINICAL TRIAL: NCT01764308
Title: Omega-3 Fatty Acid Supplementation in Acne Patients
Brief Title: Effects of Omega-3 Fatty Acid Supplementation in Acne Patients
Acronym: Omega-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient staff to complete recruitment
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Christina Kim, MD, Physician, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: O3FA
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Acne
Keywords: acne; omega-3; isotretinoin; placebo
MeSH Terms: conditions — Acne Vulgaris | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3; alpha-Linolenic Acid; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- O3FA (Experimental): Omega 3 Fatty Acid 1200mg twice a day for 24 weeks
  Interventions: Dietary Supplement: Omega-3; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): 4 tablets twice a day for 24 weeks
  Interventions: Dietary Supplement: Omega-3; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — 1200mg twice a day for 24 weeks
  Other Names: Omega-3 fatty acid; fish oil supplement; alpha-linolenic acid
Dietary Supplement: Placebo — 4 tablets twice a day for 24 weeks
  Other Names: Sugar pill

SUMMARY:
60 patients receiving isotretinoin will be recruited from the UCLA acne specialty clinic. Subjects will be randomized in a 1:1 ratio to receive placebo or omega-3 1200mg twice a day for 24 weeks.

DETAILED DESCRIPTION:
Experimental Design

60 patients receiving isotretinoin will be recruited from the UCLA acne specialty clinic. Subjects will be randomized in a 1:1 ratio to receive placebo or omega-3 1200mg twice a day for 24 weeks.

Inclusion Criteria:

* Male or female above 18 years of age.
* Moderate to severe disease at the baseline of the study identified by their dermatologist.
* Will start treatment with systemic therapy for acne in the form of either isotretinoin or oral antibiotics.
* Patients able and willing to comply with the procedures in the study protocol.

Exclusion Criteria:

* Patients with history of taking omega-3 supplements for high triglyceride levels.
* Patients taking medications for dyslipidemia, blood thinners, or high blood pressure medication.
* Patients with a history of adverse reaction to omega-3 fatty acid supplementation.
* Unwilling to give inform consent

First Visit (Baseline)

All patients will complete an intake survey. This survey will include self-assessment via Leed's standardized photo scale, and the Skindex 16 quality of life questionnaire.

Physicians will complete acne assessment on all patients. This includes lesion counts, standardized Leed's photo scale and global assessment scale 0-5.

Fasting blood sample will be obtained for chemistry and lipid panel if being treated with isotretinoin, as is standard for this therapy.

Follow-up visits at weeks 8, 16, 24:

Patients will come in at weeks 8, 16 and 24 for the following procedures:

All patients will fill out follow-up survey at each visit. The survey will elicit information regarding compliance with medication, compliance with supplementation, side effects of supplementation, side effects of acne therapy, and satisfaction with therapy.

Follow-up surveys will include patient self assessment with Leed's photo scale, and Skindex 16 questionnaire.

Physicians will complete acne assessment on all patients. This includes lesion counts, photo scale and global assessment (Grade 0-5). See attached "Physician checklist."

Patients will have fasting blood drawn for lipid panel if being treated with isotretinoin, as is standard for this therapy.

Data analysis:

In all study patients being treated for acne, lesion counts will be assessed and evaluated for any differences between patients on omega-3 fatty acid supplementation and not on supplementation.

Global assessment, photo scale assessment and Skindex-16 quality of life assessment will be compared between patients with and without supplementation.

We will compare triglyceride levels in patients being treated with isotretinoin with and without omega-3 fatty acid supplementation.

Overall satisfaction with therapy will be compared between patients with O3FA supplementation and without supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female above 18 years of age.
* Moderate to severe disease at the baseline of the study identified by their dermatologist.
* Will start treatment with systemic therapy for acne in the form of either isotretinoin or oral antibiotics.
* Patients able and willing to comply with the procedures in the study protocol.

Exclusion Criteria:

* Patients with history of taking omega-3 supplements for high triglyceride levels.
* Patients taking medications for dyslipidemia, blood thinners, or high blood pressure medication.
* Patients with a history of adverse reaction to omega-3 fatty acid supplementation.
* Unwilling to give inform consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Acne Lesion Count | up to 24 weeks
  In all study patients being treated for acne, lesion counts will be assessed and evaluated for any differences between patients on omega-3 fatty acid supplementation and not on supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Christina N Kim, MD, Principal Investigator — Kaiser Permanente; Carolyn Goh, MD, Study Chair — UCLA Division of Dermatology
Locations (1):
- University of Califonia, Los Angeles Division of Dermatology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided